CLINICAL TRIAL: NCT02474069
Title: A Randomized, Double-blind, Multicenter Study to Assess the Efficacy and Safety of 16 Weeks Secukinumab Dosage Interval Shortening in Comparison to Continued Standard Treatment (4-weekly 300 mg s.c.) in Patients With Moderate-severe Plaque Type Psoriasis Who Achieved Less Than Almost Clear Skin After 16 Weeks Under the Standard Dose of Secukinumab
Brief Title: Secukinumab Dosage Optimisation in Partial Responders With Moderate to Severe Plaque-type Psoriasis
Acronym: GAIN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAIN457ADE04; 2014-001974-32 (EudraCT Number)
Record Dates: First submitted 2015-02-26; First posted 2015-06-17 (Estimated); Results first posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-04

CONDITIONS: Moderate to Severe Plaque-type Psoriasis
Keywords: skin condition; skin disease; itching condition; psoriasis vulgaris; relapsing psoriasis; remitting psoriasis; immune-mediated systemic disease; skin lesions, red skin lesions; scaly patches; papules, plaques; itching; auto-immune; plaque-type psoriasis; plaque
MeSH Terms: conditions — Skin Diseases; Plaque, Amyloid; Pruritus | interventions — secukinumab

STUDY DESIGN:
Intervention Model Description: This was a multicenter, double-blind, randomized study in 772 patients with moderate to severe chronic plaque-type psoriasis. Patients were enrolled at 89 study sites in Germany. The study was divided into 3 phases: screening, selection phase (SP), and comparative dosing phase (CDP). In the screening phase, inclusion and exclusion criteria were confirmed. Eligible patients rolled over into a selection phase (SP) where all patients received 300 mg s.c. open-label secukinumab at baseline, Weeks 1, 2, 3, 4, 8, and 12. At Week 16, PASI response was assessed as a basis for further treatment: 300 mg s.c. secukinumab treatment every 4 weeks vesus 300 mg s.c. secukinumab treatment every 2 weeks.
  Patients who achieved at least clear or almost clear skin (≥ PASI 90) at Week 16 discontinued the study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Secukinumab Interval Shortening (Active Comparator)
  Interventions: Drug: Secukinumab
- Secukinumab 4-weekly (Active Comparator)
  Interventions: Drug: Secukinumab

INTERVENTIONS:
Drug: Secukinumab

SUMMARY:
This study is designed to support the optimal use of secukinumab by providing data to refine guidance on dosing flexibility in patients with psoriasis. The purpose of the study is to explore the effects of dosage interval shorteng to achieve PASI 90 at week 32 for patients who had less than almost clear skin at week 16.

ELIGIBILITY:
Inclusion Criteria:

Subjects eligible for inclusion in this study must fulfill all of the following criteria:

1. Subjects must be able to understand and communicate with the investigator and must give a written, signed and dated informed consent before any study related activity is performed and who are willing and capable to comply with all study procedures.
2. Men or women at least 18 years of age at time of screening.
3. Chronic plaque type psoriasis diagnosed for at least 6 months prior to baseline
4. Moderate to severe plaque type psoriasis at baseline derived from the European consensus (Mrowietz et al., 2011): BSA (Body Surface Area) >10% and PASI>10 and DLQI>10.
5. Candidates for biologic therapy who failed to respond to, or who had a contraindication to or were intolerant to previous conventional systemic therapies.
6. According to local guidelines, to exclude chest infection before initiation of a biologic immunomodulating therapy, it is necessary to have obtained an image of the chest (X-ray, computerized tomography or magnetic resonance imaging) within 12 weeks prior to screening and have this evaluated by a qualified physician.

Exclusion Criteria:

1. Forms of psoriasis other than chronic plaque-type (e.g., pustular, erythrodermic and guttata psoriasis).
2. Drug-induced psoriasis (i.e., new onset or current exacerbation from beta-blockers, calcium channel inhibitors or lithium).
3. Ongoing use of prohibited psoriasis and non-psoriasis treatments. Washout periods have to be adhered to.
4. Subjects not willing to limit UV light exposure (e.g., sunbathing and/or the use of tanning devices) during the course of the study.
5. Use of other investigational drugs at the time of enrollment, or within 30 days or 5 half-lives of enrollment, whichever is longer.
6. Previous exposure to secukinumab (AIN457) or any other biologic drug directly targeting IL-17A or the IL-17A receptor (e.g. brodalumab, ixekizumab).
7. History of hypersensitivity to any of the study drugs or to drugs with similar chemical structures.
8. Study personnel or first degree relatives of investigator(s) must not be included in the study.
9. Women who are pregnant or breast feeding (pregnancy defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (> 5 mIU/ml)) who are menstruating and capable of becoming pregnant* and not practicing a medically approved method of contraception (Pearl Index <1**) during and up to at least 4 weeks after the end of treatment. A negative pregnancy test (serum) for all women and for girls entering menarche is required with sufficient lead time before inclusion

   *definition of post-menopausal: 12 months of natural (spontaneous) amenorrhea or 6 months of spontaneous amenorrhea with serum FSH levels >40 mIU/m or 6 weeks post- surgical bilateral oophorectomy with or without hysterectomy

   **examples of particularly reliable methods with Pearl Index (PI) <1, according to guidelines of Deutsche Gesellschaft für Gynakologie und Geburtshilfe:
   * hormonal oral contraception (Combination of estrogen and gestagen, PI=0.1-0.9) hormonal vaginal ring (combination of estrogen and gestagen, PI=0.65 uncorr.; 0.4 corr.)
   * hormonal transdermal patch (combination of estrogen and gestagen, PI= 0.72 uncorr.; 0.9 corr.)
   * Estrogen-free ovulation inhibitors containing desogestrel (PI=0.14)
   * Implanted hormones containing etonogestrel (PI=0-0.08)
   * Injectable 3-month depot progestins (PI=0.3-1.4; 0.88 corr.)
   * Intra-uterine progestine device (synthetic progestin containing IUDs,PI=0.16)
   * Oral contraceptives without estrogen (e.g. "mini-pills"), nonsynthetic progesterone only IUDs, female condoms, cervical shield, periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
10. Active ongoing inflammatory diseases other than psoriasis that might confound the evaluation of the benefit of secukinumab therapy. Patients with psoriatic arthritis are not excluded.
11. Underlying condition (including, but not limited to metabolic, hematologic, renal, hepatic, pulmonary, neurologic, endocrine, cardiac, infectious or gastrointestinal) which in the opinion of the investigator significantly immunocompromises the subject and/or places the subject at unacceptable risk for receiving an immunomodulatory therapy.
12. Subjects with preexisting or recent-onset central or peripheral nervous system demyelinating disorders at discretion of the investigator.
13. Significant medical problems, including but not limited to the following: uncontrolled hypertension (≥160 systolic and/or 95 diastolic mmHg), congestive heart failure [New York Heart Association status of class III or IV].
14. Subjects with a serum creatinine level exceeding 2.0 mg/dl (176.8μmol/l) at screening.
15. Screening total white blood cell (WBC) count <2,500/μl, or platelets <100,000/μl or neutrophils <1,500/μl or hemoglobin <8.5 g/dl.
16. Active systemic infections during the last two weeks (exception: common cold) prior to screening or any infection that reoccurs on a regular basis.
17. History of an ongoing, chronic or recurrent infectious disease including recurrent respiratory and/or urinary tract infections or evidence of tuberculosis infection as defined by a positive QuantiFERON TB-Gold test at screening. Subjects with a positive or indeterminate QuantiFERON TB-Gold test may participate in the study if further full tuberculosis work up (according to local practice/guidelines) completed at least 12 weeks prior to first study drug administration establishes conclusively that the subject has no evidence of active tuberculosis. If presence of latent tuberculosis is established, then treatment must have been initiated and maintained according to local country guidelines for at least 4 weeks prior to screening.
18. Past medical history record of infection with human immunodeficiency virus (HIV), hepatitis B or hepatitis C prior to screening.
19. History of lymphoproliferative disease or any known malignancy or history of malignancy of any organ system within the past 5 years (except for skin Bowen's disease, or basal cell carcinoma or actinic keratoses that have been treated with no evidence of recurrence in the past 12 weeks; carcinoma in situ of the cervix or non-invasive malignant colon polyps that have been removed).
20. Current severe progressive or uncontrolled disease which in the judgment of the clinical investigator renders the subject unsuitable for the trial or puts the subject at increased risk.
21. Inability or unwillingness to undergo repeated venipuncture (e.g. because of poor tolerability or lack of access to veins).
22. Any medical or psychiatric condition which, in the investigator's opinion, would preclude the participant from adhering to the protocol or completing the study per protocol.
23. History or evidence of ongoing alcohol or drug abuse, within the last six months before screening.
24. Plans for administration of live vaccines during the study period or 6 weeks prior to screening.

No additional exclusions may be applied by the investigator, in order to ensure that the study population will be representative of all eligible subjects.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 772 (Actual)
Dates: Start 2015-02-08 (Actual); Primary Completion 2016-09-15 (Actual); Study Completion 2016-09-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (66):
- Germany (66):
  - Novartis Investigative Site, Bad Bentheim
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bielefeld
  - Novartis Investigative Site, Blaubeuren Abbey
  - Novartis Investigative Site, Blaustein
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Borna
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Darmstadt
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Duisburg
  - Novartis Investigative Site, Dülmen
  - Novartis Investigative Site, Düren
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Freising
  - Novartis Investigative Site, Friedrichshafen
  - Novartis Investigative Site, Garching
  - Novartis Investigative Site, Germering
  - Novartis Investigative Site, Giessen
  - Novartis Investigative Site, Glückstadt
  - Novartis Investigative Site, Goslar
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Greifswald
  - Novartis Investigative Site, Halle
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Hildesheim
  - Novartis Investigative Site, Ibbenbuehren
  - Novartis Investigative Site, Ibbenbueren
  - Novartis Investigative Site, Itzehoe
  - Novartis Investigative Site, Jena
  - Novartis Investigative Site, Kassel
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Langenau
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Lingen
  - Novartis Investigative Site, Löhne
  - Novartis Investigative Site, Lüdenscheid
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Oberhausen
  - Novartis Investigative Site, Osnabrück
  - Novartis Investigative Site, Pommelsbrunn
  - Novartis Investigative Site, Potsdam
  - Novartis Investigative Site, Quedlinburg
  - Novartis Investigative Site, Remscheid
  - Novartis Investigative Site, Rheinbach
  - Novartis Investigative Site, Schweinfurt
  - Novartis Investigative Site, Soest
  - Novartis Investigative Site, Stade
  - Novartis Investigative Site, Straubing
  - Novartis Investigative Site, Stuttgart
  - Novartis Investigative Site, Stuttgart-Weilimdorf
  - Novartis Investigative Site, Tübingen
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Weißenfels
  - Novartis Investigative Site, Wiesbaden
  - Novartis Investigative Site, Wolfenbüttel
  - Novartis Investigative Site, Wuppertal
  - Novartis Investigative Site, Würzburg

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 860 screened (not shown here). In selection phase (SP), 772 received 300 mg s.c. open-label secukinumab at baseline to wk 12. Those who did not achieve ≥Psoriasis Area and Severity Index (PASI) 75 at wk 16 discontinued. Those who had ≤ clear or almost clear skin (≥PASI75 but not PASI90) rolled over into double blind comparative dosing phase (CDP).
Pre-assignment Details: and randomized 1:1 to: a.standard treatment: 300 mg s.c. secukinumab treatment every 4 weeks (weeks 16, 20, 24, & 28) and, to maintain the blind, placebo every 4 weeks b. OR dosage interval shortening: 300 mg s.c. secukinumab treatment every 2 weeks Those who achieved at least clear or almost clear skin (≥ PASI 90) at week 16 discontinued study
Groups:
- SP - Secukinumab 300 mg s.c. (4-weekly): In the SP, all patients were treated with open-label secukinumab 300 mg s.c. at baseline, Weeks 1, 2, 3, 4, 8, and 12.
- CDP - Secukinumab 300 mg s.c. (4-weekly): In the CDP, patients received 300 mg s.c. secukinumab treatment every 4 weeks (Week 16, 20, 24, and 28) and placebo every 4 weeks (at Week 18, 22, 26 and 30).
- CDP - Secukinumab 300 mg s.c. (2-weekly): In the CDP, patients received 300 mg s.c. secukinumab treatment every 2 weeks (at weeks 16, 18, 20, 22, 24, 26, 28 and 30)
Period: Selection Phase (SP)
Arm/Group | SP - Secukinumab 300 mg s.c. (4-weekly) | CDP - Secukinumab 300 mg s.c. (4-weekly) | CDP - Secukinumab 300 mg s.c. (2-weekly)
Started | 772 | 0 | 0
Completed | 749 | 0 | 0
Not Completed | 23 | 0 | 0
Not completed — Adverse Event | 8 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — Lost to Follow-up | 4 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — No longer requires treatment | 1 | 0 | 0
Not completed — Technical Problem | 1 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 0
Not completed — Withdrawal of Informed Consent | 3 | 0 | 0
Period: Comparative Dosing Phase (CDP)
Arm/Group | SP - Secukinumab 300 mg s.c. (4-weekly) | CDP - Secukinumab 300 mg s.c. (4-weekly) | CDP - Secukinumab 300 mg s.c. (2-weekly)
Started | 0 | 162 | 163
Completed | 0 | 153 | 157
Not Completed | 0 | 9 | 6
Not completed — Adverse Event | 0 | 3 | 2
Not completed — Lost to Follow-up | 0 | 4 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Withdrawal of informed Consent | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- SP - Secukinumab 300 mg s.c. (4-weekly: In the SP, all patients were treated with open-label secukinumab 300 mg s.c. at baseline, Weeks 1, 2, 3, 4, 8, and 12. At Week 16
Arm/Group | SP - Secukinumab 300 mg s.c. (4-weekly
Number analyzed (Participants) | 772
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.8 (13.72)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 222
  Male | 550

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With PASI 90 Response at Week 32
Description: Number of participants with at least 90% improvement from baseline. PASI is a combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72 (maximal disease). Body is divided into 4 areas for scoring (head, arms, trunk, legs; each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, erythema, induration and desquamation; scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area* area score weight of section (head: 0.1, arms: 0.2 body: 0.3 legs: 0.4).
Time Frame: at 32 weeks
Population: Full Analysis Set (FAS) - Comparative Dosing Phase (CDP): consisted of all patients who were randomized and received at least one dose of study drug during the CDP and had at least one post-randomization assessment. Patients with missing PASI at week 32 were counted as non-responders, unless they were responders already at their last reported PASI.
Measure: Number; unit: participants
Arm/Group | CDP - Secukinumab 300 mg s.c. (4-weekly) | CDP - Secukinumab 300 mg s.c. (2-weekly)
Number analyzed (Participants) | 162 | 163
participants | 93 | 105
Statistical Analysis 1: Comparison: CDP - Secukinumab 300 mg s.c. (4-weekly) vs CDP - Secukinumab 300 mg s.c. (2-weekly); Logistic regression model: Logit (proportion) = treatment + PASI Score at baseline + PASI score at randomization + error; Test type: Superiority or Other; p = 0.087, ANCOVA; Odds Ratio (OR) = 0.64, 95% CI 2-sided [0.39 to 1.07]

2. Primary Outcome: Number of Participants With PASI 90 Response at Week 32 for PPS
Description: as for outcome 1
Time Frame: at week 32
Population: PPS: consisted of all patients from the FAS-CDP who completed the study without any major protocol deviation.
Measure: Number; unit: participants
Arm/Group | CDP - Secukinumab 300 mg s.c. (4-weekly) | CDP - Secukinumab 300 mg s.c. (2-weekly)
Number analyzed (Participants) | 136 | 134
participants | 81 | 85
Statistical Analysis 1: Comparison: CDP - Secukinumab 300 mg s.c. (4-weekly) vs CDP - Secukinumab 300 mg s.c. (2-weekly); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.281, ANCOVA; Odds Ratio (OR) = 0.74, 95% CI 2-sided [0.43 to 1.28]

3. Secondary Outcome: Selection Phase: Number of Participants Achieving (Psoriasis Area and Severity Index Score)PASI 50, 75, 90, 100
Description: Number of participants with at least 50, 75, 90 or 100% improvement from baseline. PASI is a combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72 (maximal disease). Body is divided into 4 areas for scoring (head, arms, trunk, legs; each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, erythema, induration and desquamation; scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area* area score weight of section (head: 0.1, arms: 0.2 body: 0.3 legs: 0.4).
Time Frame: at weeks 1, 2, 3, 4, 8, 12 and 16
Population: FAS-SP: consists of all patients that received at least one dose of study drug during the selection phase and had at least one post-baseline assessment.
Measure: Number; unit: Number of participants
Arm/Group | SP - Secukinumab 300 mg s.c. (4-weekly)
Number analyzed (Participants) | 772
Number of participants
  Week 1, PASI 50: number analyzed (Participants) | 768
  Week 1, PASI 50 | 43
  Week 1, PASI 75: number analyzed (Participants) | 768
  Week 1, PASI 75 | 3
  Week 1, PASI 90: number analyzed (Participants) | 768
  Week 1, PASI 90 | 0
  Week 1, PASI 100: number analyzed (Participants) | 768
  Week 1, PASI 100 | 0
  Week 2, PASI 50: number analyzed (Participants) | 766
  Week 2, PASI 50 | 232
  week 2, PASI 75: number analyzed (Participants) | 766
  week 2, PASI 75 | 25
  Week 2, PASI 90: number analyzed (Participants) | 766
  Week 2, PASI 90 | 5
  Week 2, PASI 100: number analyzed (Participants) | 766
  Week 2, PASI 100 | 1
  Week 3, PASI 50: number analyzed (Participants) | 766
  Week 3, PASI 50 | 468
  Week 3, PASI 75: number analyzed (Participants) | 766
  Week 3, PASI 75 | 128
  Week 3, PASI 90: number analyzed (Participants) | 766
  Week 3, PASI 90 | 22
  Week 3, PASI 100: number analyzed (Participants) | 766
  Week 3, PASI 100 | 3
  Week 4, PASI 50: number analyzed (Participants) | 768
  Week 4, PASI 50 | 591
  Week 4, PASI 75: number analyzed (Participants) | 768
  Week 4, PASI 75 | 281
  Week 4, PASI 90: number analyzed (Participants) | 768
  Week 4, PASI 90 | 71
  Week 4, PASI 100: number analyzed (Participants) | 768
  Week 4, PASI 100 | 12
  Week 8, PASI 50: number analyzed (Participants) | 762
  Week 8, PASI 50 | 718
  Week 8, PASI 75: number analyzed (Participants) | 762
  Week 8, PASI 75 | 538
  Week 8, PASI 90: number analyzed (Participants) | 762
  Week 8, PASI 90 | 266
  Week 8, PASI 100: number analyzed (Participants) | 762
  Week 8, PASI 100 | 70
  Week 12, PASI 50: number analyzed (Participants) | 761
  Week 12, PASI 50 | 733
  Week 12, PASI 75: number analyzed (Participants) | 761
  Week 12, PASI 75 | 611
  Week 12, PASI 90: number analyzed (Participants) | 761
  Week 12, PASI 90 | 370
  Week 12, PASI 100: number analyzed (Participants) | 761
  Week 12, PASI 100 | 110
  Week 16, PASI 50: number analyzed (Participants) | 753
  Week 16, PASI 50 | 732
  Week 16, PASI 75: number analyzed (Participants) | 753
  Week 16, PASI 75 | 698
  Week 16, PASI 90: number analyzed (Participants) | 753
  Week 16, PASI 90 | 363
  Week 16, PASI 100: number analyzed (Participants) | 753
  Week 16, PASI 100 | 124

4. Secondary Outcome: Comparative Dose Phase: Number of Participants Achieving Psoriasis Area and Severity Index Score (PASI) 90 and 100
Description: Number of participants with at least 90 or 100% improvement from baseline. PASI is a combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72 (maximal disease). Body is divided into 4 areas for scoring (head, arms, trunk, legs; each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, erythema, induration and desquamation; scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area* area score weight of section (head: 0.1, arms: 0.2 body: 0.3 legs: 0.4).
Time Frame: at weeks 18, 22, 30, 32
Population: FAS-CDP: consists of all patients that were randomized and received at least one dose of study drug during the comparative dosing phase and had at least one post-randomization assessment.
Measure: Number; unit: Number of participants
Arm/Group | CDP - Secukinumab 300 mg s.c. (4-weekly) | CDP - Secukinumab 300 mg s.c. (2-weekly)
Number analyzed (Participants) | 162 | 163
Number of participants
  Week 18, PASI 90 | 42 | 36
  Week 18, PASI 100 | 1 | 1
  Week 22, PASI 90 | 70 | 67
  Week 22, PASI 100 | 9 | 9
  Week 26, PASI 90 | 85 | 94
  Week 26, PASI 100 | 9 | 14
  Week 30, PASI 90 | 93 | 104
  Week 30, PASI 100 | 17 | 19
  Week 32, PASI 90 | 93 | 105
  Week 32, PASI 100 | 22 | 26

5. Secondary Outcome: Selection Phase:Summary of PASI Total Score
Description: PASI is a combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72 (maximal disease). Body is divided into 4 areas for scoring (head, arms, trunk, legs; each area is scored by itself and scores are combined for final PASI. For each area, percent of skin involved is estimated: 0 (0%) to 6 (90-100%), and severity is estimated by clinical signs, erythema, induration and desquamation; scale 0 (none) to 4 (maximum). Final PASI = sum of severity parameters for each area* area score weight of section (head: 0.1, arms: 0.2 body: 0.3 legs: 0.4).
Time Frame: at weeks 1,2,3,4,8, 12, 16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | SP - Secukinumab 300 mg s.c. (4-weekly)
Number analyzed (Participants) | 772
Score on a Scale
  week 1: number analyzed (Participants) | 768
  week 1 | 18.78 (9.629)
  week 2: number analyzed (Participants) | 766
  week 2 | 14.32 (8.435)
  week 3: number analyzed (Participants) | 766
  week 3 | 10.69 (7.372)
  week 4: number analyzed (Participants) | 768
  week 4 | 8.12 (6.494)
  week 8: number analyzed (Participants) | 762
  week 8 | 4.41 (4.544)
  Week 12: number analyzed (Participants) | 761
  Week 12 | 3.34 (3.833)
  Week 16: number analyzed (Participants) | 753
  Week 16 | 2.90 (3.816)

6. Secondary Outcome: Comparative Dose Phase: Summary of PASI Total Score
Description: as for outcome 5
Time Frame: Weeks 18, 22, 26, 30 and 32
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | CDP - Secukinumab 300 mg s.c. (4-weekly) | CDP - Secukinumab 300 mg s.c. (2-weekly)
Number analyzed (Participants) | 162 | 163
Score on a Scale
  Week 18 | 3.71 (2.532) | 3.59 (2.595)
  Week 22: number analyzed (Participants) | 161 | 161
  Week 22 | 3.24 (2.947) | 3.07 (2.726)
  Week 26: number analyzed (Participants) | 156 | 160
  Week 26 | 2.85 (2.852) | 2.68 (3.393)
  Week 30: number analyzed (Participants) | 154 | 158
  Week 30 | 2.83 (3.339) | 2.34 (2.812)
  Week 32: number analyzed (Participants) | 153 | 152
  Week 32 | 2.84 (3.552) | 2.11 (2.701)

7. Secondary Outcome: Number of Patients Achieving Dermatology Life Quality Index (DLQI) Scores of 0 or 1 by Visits in the CDP
Description: The DLQI is a ten item general dermatology disability index designed to assess health-related quality of life in adult participants with skin diseases such as eczema, psoriasis, acne and viral worts. It is a self-administered questionnaire which includes domains of daily activity, leisure, personal relationships, symptoms and feelings, treatment and school/work activities. Each domain has 4 response categories ranging from 0 (not at all) to 3 (very much). "Not relevant" is a valid score also and is scored as 0. The DLQI total score is a sum of all 10 responses. Scores range from 0 to 30 with higher scores indicating greater health-related quality of life impairment.
  The DLQI was designed to assess health-related quality of life (HRQoL) in adult patients with skin diseases including psoriasis.
Time Frame: Weeks 4, 16, 18, 22, 26, 30, 32
Population: as for outcome 4
Measure: Number; unit: participants with DLQI score 0/1
Groups:
- Secukinumab 300 mg s.c. (4-weekly): Patients received 300 mg s.c. secukinumab treatment every 4 weeks and placebo every 4 weeks
Arm/Group | Secukinumab 300 mg s.c. (4-weekly) | CDP - Secukinumab 300 mg s.c. (2-weekly)
Number analyzed (Participants) | 162 | 163
participants with DLQI score 0/1
  Week 18 | 65 | 58
  Week 22 | 70 | 73
  Week 26 | 69 | 83
  Week 30 | 75 | 89
  Week 32 | 82 | 96

8. Secondary Outcome: Number of Patients Achieving DLQI Total Score <= 5 in the CDP
Description: The DLQI is a ten item general dermatology disability index designed to assess health-related quality of life in adult participants with skin diseases such as eczema, psoriasis, acne and viral worts. It is a self-administered questionnaire which includes domains of daily activity, leisure, personal relationships, symptoms and feelings, treatment and school/work activities. Each domain has 4 response categories ranging from 0 (not at all) to 3 (very much). "Not relevant" is a valid score also and is scored as 0. The DLQI total score is a sum of all 10 responses. Scores range from 0 to 30 with higher scores indicating greater health-related quality of life impairment.
Time Frame: Weeks 4, 16, 18, 22, 26, 30, 32
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Secukinumab 300 mg s.c. (4-weekly) | CDP - Secukinumab 300 mg s.c. (2-weekly)
Number analyzed (Participants) | 162 | 163
participants
  Week 18 | 109 | 108
  Week 22 | 112 | 117
  Week 26 | 116 | 121
  Week 30 | 114 | 127
  Week 32 | 117 | 126

9. Secondary Outcome: Selection Phase: Number of Patients Achieving Investigator Global Assessment (IGA) 0 or 1
Description: The IGA scale is static, i.e. it referred exclusively to the participant's disease at the time of the assessment, and did not compare with any of the participant's previous disease states at previous visits. The scores are: 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate, 4 = severe and 5 = very severe.
Time Frame: Weeks 4, 16
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | SP - Secukinumab 300 mg s.c. (4-weekly)
Number analyzed (Participants) | 772
Participants
  week 4: number analyzed (Participants) | 768
  week 4 | 150
  week 16: number analyzed (Participants) | 759
  week 16 | 446

10. Secondary Outcome: Comparative Dose Phase: Number of Patients Achieving Investigator Global Assessment (IGA) 0 or 1
Description: as for outcome 9
Time Frame: Weeks 18, 22, 26, 30, 32
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | CDP - Secukinumab 300 mg s.c. (4-weekly) | CDP - Secukinumab 300 mg s.c. (2-weekly)
Number analyzed (Participants) | 162 | 163
Participants
  week 18 | 67 | 68
  week 22: number analyzed (Participants) | 161 | 161
  week 22 | 88 | 90
  week 26: number analyzed (Participants) | 156 | 160
  week 26 | 87 | 111
  week 30: number analyzed (Participants) | 154 | 158
  week 30 | 97 | 106
  week 32: number analyzed (Participants) | 153 | 152
  week 32 | 98 | 111

11. Secondary Outcome: Selection Phase: Summary of IGA Score
Description: as for outcome 9
Time Frame: Weeks 4, 16
Population: FAS-CDPFAS-SP: consists of all patients that received at least one dose of study drug during the selection phase and had at least one post-baseline assessment.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | SP - Secukinumab 300 mg s.c. (4-weekly)
Number analyzed (Participants) | 772
Score on a scale
  Week 4: number analyzed (Participants) | 768
  Week 4 | 2.10 (0.790)
  Week 16: number analyzed (Participants) | 759
  Week 16 | 1.26 (0.875)

12. Secondary Outcome: Comparative Dose Phase:Summary of IGA Score
Description: as for outcome 9
Time Frame: Weeks 18, 22, 26, 30, 32
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | CDP - Secukinumab 300 mg s.c. (4-weekly) | CDP - Secukinumab 300 mg s.c. (2-weekly)
Number analyzed (Participants) | 162 | 163
Score on a scale
  Week 18 | 1.63 (0.619) | 1.64 (0.656)
  Week 22: number analyzed (Participants) | 161 | 161
  Week 22 | 1.46 (0.733) | 1.42 (0.704)
  Week 26: number analyzed (Participants) | 156 | 160
  Week 26 | 1.48 (0.758) | 1.30 (0.759)
  Week 30: number analyzed (Participants) | 154 | 158
  Week 30 | 1.33 (0.848) | 1.27 (0.803)
  Week 32: number analyzed (Participants) | 153 | 152
  Week 32 | 1.30 (0.925) | 1.13 (0.819)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All AEs reported in this record are from date of First Patient First Treatment until Last Patient Last Visit) up to approximately 1 year and 4 months.
Groups:
- SP-Secukinumab: AIN457 300 mg s.c. (4-weekly): In the SP, all patients were treated with open-label secukinumab 300 mg s.c. at baseline, Weeks 1, 2, 3, 4, 8, and 12.
- CDP-Secukinumab: AIN457 300 mg s.c. (4-weekly): In the CDP, patients received 300 mg s.c. secukinumab treatment every 4 weeks (Week 16, 20, 24, and 28) and placebo every 4 weeks (at Week 18, 22, 26 and 30).
- CDP-Secukinumab: AIN457 300 mg s.c. (2-weekly): In the CDP, patients received 300 mg s.c. secukinumab treatment every 2 weeks (at weeks 16, 18, 20, 22, 24, 26, 28 and 30)
Arm/Group | SP-Secukinumab: AIN457 300 mg s.c. (4-weekly) | CDP-Secukinumab: AIN457 300 mg s.c. (4-weekly) | CDP-Secukinumab: AIN457 300 mg s.c. (2-weekly)
Serious Adverse Events (participants affected / at risk) | 32/772 | 8/162 | 4/163
Other Adverse Events (participants affected / at risk) | 510/772 | 85/162 | 87/163
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SP-Secukinumab: AIN457 300 mg s.c. (4-weekly) (N=772) | CDP-Secukinumab: AIN457 300 mg s.c. (4-weekly) (N=162) | CDP-Secukinumab: AIN457 300 mg s.c. (2-weekly) (N=163)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 0 | 0
CARDIAC FAILURE (Cardiac disorders) | 1 | 0 | 0
MYOCARDITIS (Cardiac disorders) | 1 | 0 | 0
VENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 1 | 0 | 0
COLITIS ULCERATIVE (Gastrointestinal disorders) | 1 | 0 | 0
DIARRHOEA (Gastrointestinal disorders) | 1 | 0 | 0
GASTRITIS (Gastrointestinal disorders) | 1 | 0 | 0
UMBILICAL HERNIA (Gastrointestinal disorders) | 1 | 0 | 0
CHEST PAIN (General disorders) | 0 | 1 | 0
CHILLS (General disorders) | 1 | 0 | 0
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 1 | 0 | 0
IMPAIRED HEALING (General disorders) | 0 | 1 | 0
BILIARY COLIC (Hepatobiliary disorders) | 1 | 0 | 0
CHOLECYSTITIS CHRONIC (Hepatobiliary disorders) | 1 | 0 | 0
ERYSIPELAS (Infections and infestations) | 0 | 1 | 0
MASTOIDITIS (Infections and infestations) | 0 | 1 | 0
PYODERMA (Infections and infestations) | 0 | 1 | 0
SINUSITIS (Infections and infestations) | 0 | 1 | 0
TONSILLITIS (Infections and infestations) | 1 | 0 | 0
VARICELLA (Infections and infestations) | 0 | 0 | 1
CHEST INJURY (Injury, poisoning and procedural complications) | 0 | 1 | 0
CONCUSSION (Injury, poisoning and procedural complications) | 1 | 0 | 0
CONTUSION (Injury, poisoning and procedural complications) | 0 | 1 | 0
FALL (Injury, poisoning and procedural complications) | 0 | 1 | 0
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 1
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1
LIGAMENT RUPTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
RADIAL HEAD DISLOCATION (Injury, poisoning and procedural complications) | 1 | 0 | 0
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 2 | 0 | 0
STERNAL FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
TENDON RUPTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
WOUND (Injury, poisoning and procedural complications) | 0 | 1 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 1 | 0
HEPATIC ENZYME INCREASED (Investigations) | 1 | 0 | 0
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
B-CELL LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
MYCOSIS FUNGOIDES (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
PANCREATIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
CEREBRAL ISCHAEMIA (Nervous system disorders) | 0 | 1 | 0
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 | 0 | 1
INTERCOSTAL NEURALGIA (Nervous system disorders) | 0 | 1 | 0
MANIA (Psychiatric disorders) | 1 | 0 | 0
PANIC ATTACK (Psychiatric disorders) | 1 | 0 | 0
FIBRILLARY GLOMERULONEPHRITIS (Renal and urinary disorders) | 1 | 0 | 0
RENAL CYST HAEMORRHAGE (Renal and urinary disorders) | 1 | 0 | 0
URETEROLITHIASIS (Renal and urinary disorders) | 1 | 0 | 0
ASTHMA EXERCISE INDUCED (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
HYPERVENTILATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
ACROKERATOSIS PARANEOPLASTICA (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
DERMATITIS EXFOLIATIVE (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
SKIN ULCER (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
HAEMORRHAGE (Vascular disorders) | 1 | 0 | 0
HYPERTENSIVE CRISIS (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 0.0001% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SP-Secukinumab: AIN457 300 mg s.c. (4-weekly) (N=772) | CDP-Secukinumab: AIN457 300 mg s.c. (4-weekly) (N=162) | CDP-Secukinumab: AIN457 300 mg s.c. (2-weekly) (N=163)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 1 | 0 | 0
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 2 | 2 | 0
LYMPHOPENIA (Blood and lymphatic system disorders) | 1 | 0 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 1 | 0 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 | 0 | 1
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 1 | 1
ATRIOVENTRICULAR BLOCK (Cardiac disorders) | 0 | 0 | 1
BUNDLE BRANCH BLOCK LEFT (Cardiac disorders) | 1 | 0 | 0
SINUS ARRHYTHMIA (Cardiac disorders) | 1 | 0 | 0
TACHYCARDIA (Cardiac disorders) | 1 | 0 | 0
CONGENITAL NAEVUS (Congenital, familial and genetic disorders) | 1 | 0 | 0
EAR PAIN (Ear and labyrinth disorders) | 1 | 2 | 0
EAR PRURITUS (Ear and labyrinth disorders) | 2 | 0 | 0
HYPOACUSIS (Ear and labyrinth disorders) | 0 | 1 | 0
SUDDEN HEARING LOSS (Ear and labyrinth disorders) | 1 | 0 | 0
TINNITUS (Ear and labyrinth disorders) | 2 | 0 | 0
TYMPANIC MEMBRANE PERFORATION (Ear and labyrinth disorders) | 1 | 0 | 0
VERTIGO (Ear and labyrinth disorders) | 3 | 0 | 0
HYPERTHYROIDISM (Endocrine disorders) | 1 | 0 | 0
HYPOTHYROIDISM (Endocrine disorders) | 0 | 0 | 1
THYROID CYST (Endocrine disorders) | 1 | 0 | 0
BLEPHARITIS (Eye disorders) | 3 | 1 | 0
CATARACT (Eye disorders) | 1 | 0 | 0
CHALAZION (Eye disorders) | 2 | 0 | 0
CONJUNCTIVAL HYPERAEMIA (Eye disorders) | 1 | 0 | 0
CONJUNCTIVITIS ALLERGIC (Eye disorders) | 4 | 1 | 1
DRY EYE (Eye disorders) | 3 | 0 | 1
ECZEMA EYELIDS (Eye disorders) | 2 | 0 | 1
EYE IRRITATION (Eye disorders) | 1 | 0 | 0
EYE PAIN (Eye disorders) | 2 | 0 | 0
EYE SWELLING (Eye disorders) | 2 | 1 | 0
EYELID OEDEMA (Eye disorders) | 1 | 0 | 1
EYELIDS PRURITUS (Eye disorders) | 1 | 0 | 0
INTRAOCULAR HAEMATOMA (Eye disorders) | 0 | 0 | 1
KERATITIS (Eye disorders) | 1 | 0 | 0
LACRIMATION INCREASED (Eye disorders) | 4 | 0 | 0
VISUAL IMPAIRMENT (Eye disorders) | 3 | 0 | 0
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 | 0 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 | 1 | 0
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 2 | 0 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 17 | 1 | 1
ANAL SKIN TAGS (Gastrointestinal disorders) | 1 | 0 | 0
ANORECTAL DISCOMFORT (Gastrointestinal disorders) | 1 | 0 | 0
APHTHOUS ULCER (Gastrointestinal disorders) | 2 | 0 | 0
COLITIS (Gastrointestinal disorders) | 2 | 0 | 0
COLITIS MICROSCOPIC (Gastrointestinal disorders) | 1 | 0 | 0
CONSTIPATION (Gastrointestinal disorders) | 2 | 0 | 0
DENTAL CARIES (Gastrointestinal disorders) | 1 | 0 | 0
DIARRHOEA (Gastrointestinal disorders) | 34 | 3 | 1
DRY MOUTH (Gastrointestinal disorders) | 4 | 0 | 0
DYSPEPSIA (Gastrointestinal disorders) | 2 | 1 | 0
DYSPHAGIA (Gastrointestinal disorders) | 2 | 0 | 0
EPULIS (Gastrointestinal disorders) | 1 | 0 | 0
FAECES SOFT (Gastrointestinal disorders) | 1 | 0 | 0
FLATULENCE (Gastrointestinal disorders) | 3 | 0 | 0
FREQUENT BOWEL MOVEMENTS (Gastrointestinal disorders) | 0 | 1 | 0
GASTRITIS (Gastrointestinal disorders) | 5 | 0 | 1
GASTRITIS EROSIVE (Gastrointestinal disorders) | 0 | 0 | 1
GASTROINTESTINAL PAIN (Gastrointestinal disorders) | 0 | 1 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 6 | 0 | 1
GINGIVAL DISORDER (Gastrointestinal disorders) | 1 | 0 | 0
GINGIVAL EROSION (Gastrointestinal disorders) | 1 | 0 | 0
HAEMORRHOIDS (Gastrointestinal disorders) | 1 | 0 | 0
HYPOAESTHESIA ORAL (Gastrointestinal disorders) | 1 | 0 | 0
INTRA-ABDOMINAL HAEMATOMA (Gastrointestinal disorders) | 1 | 0 | 0
LARGE INTESTINE POLYP (Gastrointestinal disorders) | 1 | 0 | 0
LIP BLISTER (Gastrointestinal disorders) | 0 | 0 | 1
LIP DRY (Gastrointestinal disorders) | 1 | 0 | 0
MALLORY-WEISS SYNDROME (Gastrointestinal disorders) | 1 | 0 | 0
MOUTH SWELLING (Gastrointestinal disorders) | 1 | 0 | 0
MOUTH ULCERATION (Gastrointestinal disorders) | 1 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 9 | 1 | 0
PARAESTHESIA ORAL (Gastrointestinal disorders) | 1 | 0 | 0
POUCHITIS (Gastrointestinal disorders) | 1 | 0 | 0
TONGUE COATED (Gastrointestinal disorders) | 1 | 0 | 0
TONGUE DISCOLOURATION (Gastrointestinal disorders) | 0 | 0 | 1
TOOTHACHE (Gastrointestinal disorders) | 9 | 0 | 0
VASCULITIS GASTROINTESTINAL (Gastrointestinal disorders) | 0 | 1 | 0
VOMITING (Gastrointestinal disorders) | 3 | 1 | 1
APPLICATION SITE HAEMATOMA (General disorders) | 1 | 0 | 0
ASTHENIA (General disorders) | 1 | 0 | 0
CHILLS (General disorders) | 1 | 0 | 0
DRUG THERAPEUTIC INCOMPATIBILITY (General disorders) | 0 | 0 | 1
FATIGUE (General disorders) | 28 | 4 | 3
FEELING HOT (General disorders) | 1 | 0 | 0
IMPAIRED HEALING (General disorders) | 1 | 0 | 0
INFLUENZA LIKE ILLNESS (General disorders) | 10 | 2 | 1
INJECTION SITE BRUISING (General disorders) | 2 | 0 | 0
INJECTION SITE ERYTHEMA (General disorders) | 1 | 0 | 0
INJECTION SITE HAEMATOMA (General disorders) | 1 | 0 | 0
INJECTION SITE HAEMORRHAGE (General disorders) | 0 | 0 | 1
INJECTION SITE PAIN (General disorders) | 3 | 0 | 1
INJECTION SITE PRURITUS (General disorders) | 2 | 0 | 0
INJURY ASSOCIATED WITH DEVICE (General disorders) | 0 | 1 | 0
NON-CARDIAC CHEST PAIN (General disorders) | 3 | 0 | 0
OEDEMA PERIPHERAL (General disorders) | 4 | 0 | 0
PERIPHERAL SWELLING (General disorders) | 1 | 0 | 1
PUNCTURE SITE REACTION (General disorders) | 1 | 0 | 0
PYREXIA (General disorders) | 9 | 0 | 0
SENSATION OF FOREIGN BODY (General disorders) | 1 | 1 | 0
THIRST (General disorders) | 1 | 0 | 0
BILIARY COLIC (Hepatobiliary disorders) | 1 | 0 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 0 | 1 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 1 | 0 | 0
HEPATIC STEATOSIS (Hepatobiliary disorders) | 3 | 0 | 0
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 1 | 1 | 0
SEASONAL ALLERGY (Immune system disorders) | 2 | 0 | 0
ABDOMINAL ABSCESS (Infections and infestations) | 1 | 0 | 0
ABSCESS (Infections and infestations) | 1 | 0 | 0
ANGULAR CHEILITIS (Infections and infestations) | 5 | 0 | 1
BACTERIAL INFECTION (Infections and infestations) | 1 | 0 | 0
BACTERIAL RHINITIS (Infections and infestations) | 0 | 1 | 0
BACTERIAL VAGINOSIS (Infections and infestations) | 0 | 2 | 0
BALANITIS CANDIDA (Infections and infestations) | 2 | 0 | 1
BODY TINEA (Infections and infestations) | 2 | 0 | 0
BRONCHITIS (Infections and infestations) | 10 | 2 | 2
BRONCHITIS BACTERIAL (Infections and infestations) | 0 | 0 | 1
BRONCHITIS VIRAL (Infections and infestations) | 0 | 0 | 1
CANDIDA INFECTION (Infections and infestations) | 5 | 0 | 0
CONJUNCTIVITIS (Infections and infestations) | 8 | 1 | 2
CONJUNCTIVITIS BACTERIAL (Infections and infestations) | 1 | 0 | 0
CYSTITIS (Infections and infestations) | 4 | 2 | 1
CYSTITIS BACTERIAL (Infections and infestations) | 0 | 0 | 1
ECZEMA IMPETIGINOUS (Infections and infestations) | 1 | 0 | 0
EPIDIDYMITIS (Infections and infestations) | 0 | 0 | 1
EPIGLOTTITIS (Infections and infestations) | 1 | 0 | 0
ERYSIPELAS (Infections and infestations) | 2 | 1 | 0
FOLLICULITIS (Infections and infestations) | 13 | 4 | 2
FUNGAL INFECTION (Infections and infestations) | 1 | 0 | 0
FUNGAL SKIN INFECTION (Infections and infestations) | 5 | 0 | 0
FURUNCLE (Infections and infestations) | 3 | 0 | 0
GASTROENTERITIS (Infections and infestations) | 7 | 1 | 0
GASTROENTERITIS VIRAL (Infections and infestations) | 1 | 0 | 0
GASTROINTESTINAL INFECTION (Infections and infestations) | 8 | 1 | 1
GASTROINTESTINAL VIRAL INFECTION (Infections and infestations) | 2 | 0 | 1
GENITAL CANDIDIASIS (Infections and infestations) | 1 | 0 | 0
GENITAL INFECTION FUNGAL (Infections and infestations) | 1 | 0 | 0
GINGIVITIS (Infections and infestations) | 4 | 1 | 0
HELICOBACTER INFECTION (Infections and infestations) | 1 | 0 | 0
HERPES SIMPLEX (Infections and infestations) | 3 | 0 | 0
HERPES VIRUS INFECTION (Infections and infestations) | 1 | 0 | 0
HERPES ZOSTER (Infections and infestations) | 2 | 2 | 0
HERPES ZOSTER INFECTION NEUROLOGICAL (Infections and infestations) | 0 | 0 | 1
HORDEOLUM (Infections and infestations) | 1 | 0 | 0
IMPETIGO (Infections and infestations) | 2 | 0 | 0
INFLUENZA (Infections and infestations) | 9 | 2 | 2
LABYRINTHITIS (Infections and infestations) | 2 | 0 | 0
LARYNGITIS (Infections and infestations) | 0 | 1 | 0
LOCALISED INFECTION (Infections and infestations) | 1 | 0 | 0
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1 | 0
LYME DISEASE (Infections and infestations) | 1 | 0 | 0
MUCOSAL INFECTION (Infections and infestations) | 1 | 0 | 0
NAIL BED INFECTION (Infections and infestations) | 1 | 0 | 0
NASOPHARYNGITIS (Infections and infestations) | 168 | 23 | 27
OESOPHAGEAL CANDIDIASIS (Infections and infestations) | 2 | 0 | 0
ORAL CANDIDIASIS (Infections and infestations) | 14 | 2 | 3
ORAL FUNGAL INFECTION (Infections and infestations) | 1 | 1 | 0
ORAL HERPES (Infections and infestations) | 15 | 1 | 1
ORCHITIS (Infections and infestations) | 1 | 0 | 0
OTITIS EXTERNA (Infections and infestations) | 4 | 1 | 1
OTITIS MEDIA (Infections and infestations) | 4 | 0 | 1
OTITIS MEDIA ACUTE (Infections and infestations) | 0 | 0 | 1
PARONYCHIA (Infections and infestations) | 2 | 0 | 1
PERICHONDRITIS (Infections and infestations) | 1 | 0 | 0
PERIODONTITIS (Infections and infestations) | 1 | 0 | 1
PHARYNGITIS (Infections and infestations) | 6 | 2 | 1
PHARYNGITIS BACTERIAL (Infections and infestations) | 1 | 0 | 0
PHARYNGITIS STREPTOCOCCAL (Infections and infestations) | 1 | 0 | 0
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 1 | 0 | 0
PULPITIS DENTAL (Infections and infestations) | 5 | 0 | 1
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0
RHINITIS (Infections and infestations) | 16 | 1 | 0
SINUSITIS (Infections and infestations) | 8 | 2 | 1
SKIN CANDIDA (Infections and infestations) | 1 | 0 | 1
SKIN INFECTION (Infections and infestations) | 2 | 0 | 1
STAPHYLOCOCCAL SKIN INFECTION (Infections and infestations) | 1 | 0 | 0
SUBCUTANEOUS ABSCESS (Infections and infestations) | 2 | 1 | 0
TINEA INFECTION (Infections and infestations) | 2 | 0 | 0
TINEA PEDIS (Infections and infestations) | 8 | 3 | 1
TONSILLITIS (Infections and infestations) | 6 | 1 | 2
TONSILLITIS BACTERIAL (Infections and infestations) | 0 | 0 | 1
TOOTH INFECTION (Infections and infestations) | 2 | 2 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 | 1 | 0
URETHRITIS (Infections and infestations) | 1 | 1 | 0
URINARY TRACT INFECTION (Infections and infestations) | 3 | 0 | 1
VIRAL INFECTION (Infections and infestations) | 1 | 1 | 1
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 | 0 | 1
VULVOVAGINAL CANDIDIASIS (Infections and infestations) | 1 | 0 | 0
VULVOVAGINAL MYCOTIC INFECTION (Infections and infestations) | 2 | 1 | 0
ACCIDENT AT WORK (Injury, poisoning and procedural complications) | 1 | 0 | 0
ANIMAL BITE (Injury, poisoning and procedural complications) | 1 | 0 | 1
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 1 | 1 | 0
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 2 | 0 | 0
ARTHROPOD STING (Injury, poisoning and procedural complications) | 3 | 0 | 0
BURN ORAL CAVITY (Injury, poisoning and procedural complications) | 1 | 0 | 0
CERVICAL VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
CONTUSION (Injury, poisoning and procedural complications) | 5 | 0 | 0
CRANIOCEREBRAL INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 0
FALL (Injury, poisoning and procedural complications) | 1 | 1 | 0
FOREIGN BODY IN EYE (Injury, poisoning and procedural complications) | 1 | 0 | 1
HAND FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 0 | 0 | 1
JOINT INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 0
LACERATION (Injury, poisoning and procedural complications) | 2 | 1 | 0
LIGAMENT RUPTURE (Injury, poisoning and procedural complications) | 2 | 0 | 0
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 6 | 0 | 0
LIMB INJURY (Injury, poisoning and procedural complications) | 2 | 0 | 0
MENISCUS INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 0
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 2 | 0 | 0
PLAQUE SHIFT (Injury, poisoning and procedural complications) | 0 | 1 | 0
PROCEDURAL DIZZINESS (Injury, poisoning and procedural complications) | 1 | 0 | 0
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 2 | 1 | 1
RIB FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 | 0 | 0
SKIN ABRASION (Injury, poisoning and procedural complications) | 3 | 0 | 0
SUBCUTANEOUS HAEMATOMA (Injury, poisoning and procedural complications) | 2 | 0 | 0
SUNBURN (Injury, poisoning and procedural complications) | 2 | 1 | 0
TENDON RUPTURE (Injury, poisoning and procedural complications) | 0 | 1 | 0
THERMAL BURN (Injury, poisoning and procedural complications) | 1 | 0 | 0
TOOTH FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1
WOUND (Injury, poisoning and procedural complications) | 2 | 0 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 3 | 1 | 1
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 2 | 0 | 0
BILIRUBIN URINE PRESENT (Investigations) | 1 | 0 | 0
BLOOD CHOLESTEROL INCREASED (Investigations) | 0 | 0 | 1
BLOOD CREATININE INCREASED (Investigations) | 0 | 1 | 0
BLOOD TRIGLYCERIDES INCREASED (Investigations) | 0 | 0 | 1
BLOOD URINE PRESENT (Investigations) | 2 | 0 | 0
BODY TEMPERATURE INCREASED (Investigations) | 1 | 0 | 0
ELECTROCARDIOGRAM ABNORMAL (Investigations) | 1 | 0 | 1
ELECTROCARDIOGRAM Q WAVE ABNORMAL (Investigations) | 1 | 0 | 0
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 3 | 0 | 0
HEPATIC ENZYME INCREASED (Investigations) | 2 | 0 | 0
HIGH DENSITY LIPOPROTEIN DECREASED (Investigations) | 0 | 0 | 1
HUMAN CHORIONIC GONADOTROPIN INCREASED (Investigations) | 1 | 0 | 0
LIVER FUNCTION TEST INCREASED (Investigations) | 1 | 0 | 0
MONOCYTE COUNT INCREASED (Investigations) | 1 | 0 | 0
NEUTROPHIL COUNT DECREASED (Investigations) | 2 | 0 | 0
PLATELET COUNT DECREASED (Investigations) | 1 | 0 | 0
TRANSAMINASES INCREASED (Investigations) | 0 | 1 | 0
WEIGHT INCREASED (Investigations) | 1 | 1 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 | 0 | 0
DIABETES MELLITUS (Metabolism and nutrition disorders) | 2 | 1 | 1
FLUID RETENTION (Metabolism and nutrition disorders) | 1 | 0 | 0
GOUT (Metabolism and nutrition disorders) | 1 | 0 | 0
HAEMOSIDEROSIS (Metabolism and nutrition disorders) | 1 | 0 | 0
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 2 | 1 | 0
HYPERKALAEMIA (Metabolism and nutrition disorders) | 2 | 0 | 0
HYPERLIPIDAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 3 | 0 | 0
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 | 1 | 0
IRON DEFICIENCY (Metabolism and nutrition disorders) | 0 | 1 | 0
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 0 | 1
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 1 | 0 | 0
ZINC DEFICIENCY (Metabolism and nutrition disorders) | 1 | 0 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 21 | 4 | 3
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 9 | 3 | 3
BURSITIS (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
FIBROMYALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
JOINT CREPITATION (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
JOINT EFFUSION (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0
METATARSALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
MUSCLE TIGHTNESS (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 4 | 1 | 0
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 12 | 0 | 0
PATELLOFEMORAL PAIN SYNDROME (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
PSORIATIC ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
RHEUMATIC DISORDER (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
SCOLIOSIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
SPINAL OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
SPINAL PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
SYNOVIAL CYST (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
TENDONITIS (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
TENOSYNOVITIS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
DYSPLASTIC NAEVUS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
FIBROMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
FIBROUS HISTIOCYTOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
MELANOCYTIC NAEVUS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
MONOCLONAL GAMMOPATHY (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
SEBORRHOEIC KERATOSIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
SKIN PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 3 | 1
BURNING SENSATION (Nervous system disorders) | 0 | 1 | 0
CARPAL TUNNEL SYNDROME (Nervous system disorders) | 0 | 1 | 0
CERVICOGENIC VERTIGO (Nervous system disorders) | 0 | 0 | 1
DIZZINESS (Nervous system disorders) | 3 | 1 | 0
DYSAESTHESIA (Nervous system disorders) | 1 | 0 | 0
DYSGEUSIA (Nervous system disorders) | 2 | 0 | 1
HEADACHE (Nervous system disorders) | 60 | 5 | 5
HYPERAESTHESIA (Nervous system disorders) | 1 | 0 | 0
MIGRAINE (Nervous system disorders) | 2 | 0 | 1
NERVE COMPRESSION (Nervous system disorders) | 0 | 1 | 0
NEURALGIA (Nervous system disorders) | 2 | 0 | 0
NEURITIS (Nervous system disorders) | 0 | 0 | 1
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 | 0 | 0
ORTHOSTATIC INTOLERANCE (Nervous system disorders) | 0 | 1 | 0
SCIATICA (Nervous system disorders) | 4 | 1 | 4
SOMNOLENCE (Nervous system disorders) | 1 | 0 | 0
ALCOHOL ABUSE (Psychiatric disorders) | 1 | 0 | 0
DEPRESSION (Psychiatric disorders) | 3 | 0 | 0
INITIAL INSOMNIA (Psychiatric disorders) | 1 | 0 | 0
INSOMNIA (Psychiatric disorders) | 1 | 0 | 0
MOOD SWINGS (Psychiatric disorders) | 1 | 0 | 0
NERVOUSNESS (Psychiatric disorders) | 1 | 0 | 0
SLEEP DISORDER (Psychiatric disorders) | 1 | 0 | 0
DYSURIA (Renal and urinary disorders) | 0 | 0 | 1
HAEMATURIA (Renal and urinary disorders) | 5 | 1 | 0
LEUKOCYTURIA (Renal and urinary disorders) | 4 | 0 | 0
NEPHROLITHIASIS (Renal and urinary disorders) | 2 | 0 | 0
POLLAKIURIA (Renal and urinary disorders) | 2 | 0 | 0
PROTEINURIA (Renal and urinary disorders) | 3 | 0 | 0
BALANOPOSTHITIS (Reproductive system and breast disorders) | 1 | 0 | 0
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 1 | 0 | 0
BREAST CYST (Reproductive system and breast disorders) | 1 | 0 | 0
DYSMENORRHOEA (Reproductive system and breast disorders) | 1 | 0 | 0
MENOPAUSAL SYMPTOMS (Reproductive system and breast disorders) | 1 | 0 | 0
MENSTRUATION IRREGULAR (Reproductive system and breast disorders) | 2 | 0 | 0
METRORRHAGIA (Reproductive system and breast disorders) | 1 | 0 | 0
PROSTATITIS (Reproductive system and breast disorders) | 0 | 0 | 1
PRURITUS GENITAL (Reproductive system and breast disorders) | 2 | 0 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 12 | 0 | 2
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
NASAL INFLAMMATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
NASAL MUCOSAL EROSION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OROPHARYNGEAL DISCOMFORT (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 12 | 1 | 2
PHARYNGEAL INFLAMMATION (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 10 | 1 | 0
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
THROAT IRRITATION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
ACNE (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
ACTINIC KERATOSIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
ALOPECIA (Skin and subcutaneous tissue disorders) | 5 | 0 | 0
ALOPECIA AREATA (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
BLISTER (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
BLOOD BLISTER (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
DERMAL CYST (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
DERMATITIS ALLERGIC (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 5 | 2 | 0
DRUG ERUPTION (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
DYSHIDROTIC ECZEMA (Skin and subcutaneous tissue disorders) | 3 | 2 | 2
ECZEMA (Skin and subcutaneous tissue disorders) | 10 | 4 | 1
ECZEMA WEEPING (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
ERYTHEMA (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
ERYTHEMA NODOSUM (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
INGROWING NAIL (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
INTERTRIGO (Skin and subcutaneous tissue disorders) | 8 | 0 | 1
MILIARIA (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
MYXOID CYST (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
PAIN OF SKIN (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
PAPULE (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
PETECHIAE (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
PHOTODERMATOSIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
PHOTOSENSITIVITY REACTION (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
PRURIGO (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 32 | 2 | 0
PRURITUS ALLERGIC (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
PRURITUS GENERALISED (Skin and subcutaneous tissue disorders) | 8 | 1 | 1
PSORIASIS (Skin and subcutaneous tissue disorders) | 3 | 2 | 2
PUSTULAR PSORIASIS (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
RASH (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
RASH MACULAR (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
RASH PAPULAR (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
ROSACEA (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
SEBORRHOEA (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
SEBORRHOEIC DERMATITIS (Skin and subcutaneous tissue disorders) | 13 | 0 | 1
SKIN ATROPHY (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
SKIN EXFOLIATION (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
SKIN FISSURES (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
SKIN IRRITATION (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
SKIN PLAQUE (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
SKIN ULCER (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
SKIN ULCER HAEMORRHAGE (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
SOLAR DERMATITIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
URTICARIA (Skin and subcutaneous tissue disorders) | 7 | 1 | 1
DIASTOLIC HYPERTENSION (Vascular disorders) | 1 | 0 | 0
FLUSHING (Vascular disorders) | 1 | 0 | 0
HAEMATOMA (Vascular disorders) | 1 | 1 | 1
HAEMORRHAGE (Vascular disorders) | 1 | 0 | 0
HYPERTENSION (Vascular disorders) | 8 | 3 | 4
LYMPHOEDEMA (Vascular disorders) | 0 | 1 | 0
PERIPHERAL VENOUS DISEASE (Vascular disorders) | 0 | 1 | 0
VARICOSE VEIN (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial